CLINICAL TRIAL: NCT06659367
Title: Institute for Cardiovascular Diseases "Dedinje" Fractional Flow Reserve (FFR) and Quantitative Flow Ratio (QFR) Registry
Brief Title: Dedinje FFR/QFR Registry
Status: Recruiting | Type: Observational
Sponsor: Institute for Cardiovascular Diseases Dedinje (Other)
Responsible Party: Principal Investigator, Natalija Odanovic, Principal Investigator, Institute for Cardiovascular Diseases Dedinje
Other Study IDs: IRB4669
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease (CAD); Fractional Flow Reserve
Keywords: coronary artery disease; fractional flow reserve; quantitative flow ratio; FFR; QFR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Quantitative Flow Ratio (QFR) has shown good diagnostic performance against Fractional Flow Reserve (FFR) in several meta-analyses, comparable or even superior to nonhyperemic pressure ratios. However, the reproducibility of QFR is modest and there is high inter- and intra-observer variability even when fairly experienced but non-core lab operators (at least 150 QFR procedure experience) are performing the analysis. Although smaller studies have demonstrated that non-core analysis and even paramedical user analysis can have good correlation with FFR, the concern about the diagnostic performance of QFR in real-world clinical practice by inexperienced users remains.

The primary objective of "Dedinje FFR/QFR Registry" is to determine the feasibility and diagnostic performance of QFR analysis by vendor-certified inexperienced medical users in a real-world setting using FFR as the gold standard. All patients >18 years old who present to the Institute for Cardiovascular Diseases "Dedinje" and undergo a planned or ad hoc FFR procedure will be asked to participate in the registry. FFR procedure is performed according to the standardized institutional protocol. QFR analysis will be subsequently performed offline according to a standard operating procedure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Had a clinically indicated FFR procedure performed (either as a planned procedure or ad hoc)

Exclusion Criteria:

* Declines to participate in the registry and provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years old who present to the Institute for Cardiovascular Diseases "Dedinje" and undergo a planned or ad hoc FFR procedure will be asked to participate in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2029-10-02 (Estimated); Study Completion 2034-10-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between Quantitative Flow Ratio (QFR) and Fractional Flow Reserve (FFR) | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  correlation coefficient (r) between Quantitative Flow Ratio (QFR) and Fractional Flow Reserve (FFR)
Sensitivity of Quantitative Flow Ratio (QFR) | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Sensitivity of Quantitative Flow Ratio (QFR) against Fractional Flow Reserve (FFR) as the gold standard
Specificity of Quantitative Flow Ratio (QFR) | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Specificity of Quantitative Flow Ratio (QFR) against Fractional Flow Reserve (FFR) as the gold standard
Positive predictive value of Quantitative Flow Ratio (QFR) | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Positive predictive value of Quantitative Flow Ratio (QFR) against Fractional Flow Reserve (FFR) as the gold standard
Negative predictive value of Quantitative Flow Ratio (QFR) | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Negative predictive value of Quantitative Flow Ratio (QFR) against Fractional Flow Reserve (FFR) as the gold standard
Diagnostic gray zone | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Quantitative Flow Ratio (QFR) limits for achieving 95% sensitivity and specificity in comparison to Fractional Flow Reserve (FFR)
Diagnostic accuracy of Quantitative Flow Ratio (QFR) against Fractional Flow Reserve (FFR) | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Area under the curve (using cutoff values of <=0.80 for both methods)

SECONDARY OUTCOMES:
Diagnostic performance of nonhyperemic pressure ratios and 3-dimensional Quantitative Coronary Angiography (3D-QCA) against Fractional Flow Reserve (FFR) as the gold standard | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Sensitivity, specificity, positive predictive value and negative predictive value of nonhyperemic pressure ratios and 3-dimensional Quantitative Coronary Angiography (3D-QCA) against Fractional Flow Reserve (FFR)
Diagnostic accuracy of nonhyperemic pressure ratios and 3-dimensional Quantitative Coronary Angiography (3D-QCA) against Fractional Flow Reserve (FFR) as the gold standard | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Area under the curve (using cutoff values of <=0.89 for nonhyperemic pressure ratios and >=50% diameter stenosis for 3-dimensional Quantitative Coronary Angiography (3D-QCA)) against Fractional Flow Reserve (FFR, cutoff value <=0.80)
Inter-observer variability | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Coefficient of variation for repeated Quantitative Flow Ratio (QFR) computation between users, standard deviation for repeated Quantitative Flow Ratio (QFR) measurements between users, binary diagnostic classification agreement between users
Intra-observer variability | at the time of Quantitative Flow Ratio (QFR) analysis completion (up to 1 year)
  Coefficient of variation for repeated Quantitative Flow Ratio (QFR) computation within users, standard deviation for repeated Quantitative Flow Ratio (QFR) measurements within users, binary diagnostic classification agreement within users
All-cause death | at 6 months, 1 year and annually for 5 years
  All-cause death
Myocardial infarction | at 6 months, 1 year and annually for 5 years
  Myocardial infarction
Vessel-oriented composite outcome | at 6 months, 1 year and annually for 5 years
  Cardiac death, vessel-related myocardial infarction and ischemia-driven target vessel revascularization
Change in Seattle Angina Questionnaire-7 Items Score (SAQ-7) at 6 months | 6 months
  Change in Seattle Angina Questionnaire-7 Items Score (SAQ-7) at 6 months from the time of the Fractional Flow Reserve (FFR) procedure. (scale 0-100, 100 = full health, 0 = worst health)
Change in EuroQol-5 Dimensions- 5 Levels (EQ-5D-5L) Score | 6 months
  Change in EuroQol-5 Dimensions- 5 Levels (EQ-5D-5L) Score at 6 months from the time of the Fractional Flow Reserve (FFR) procedure (scale 5-25, 5= no problems in any dimension, 25= extreme problems on all dimensions; visual analogue scale 0-100, 0= worst health possible, 100= best health possible)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Cardiovascular Diseases "Dedinje", Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
IPD contains sensitive identifying patient information that patients are told will not be shared with anyone outside of the primary team of researchers.